CLINICAL TRIAL: NCT07389109
Title: A Long-term Safety and Efficacy Study of N-Acetyl-GED-0507-34-LEVO Gel 5%, in Subjects With Acne Vulgaris (GEDACNE-LT)
Acronym: GEDACNE-LT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PPM Services S.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAC-GED-0507-ACN-01-23-LT; 2023-510342-24-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-12; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-10

CONDITIONS: Acne Vulgaris
Keywords: acne; acne vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N-Acetyl-GED-0507-34-Levo 5% gel (Experimental)
  Interventions: Drug: N-Acetyl-GED-0507-34-LEVO gel 5%

INTERVENTIONS:
Drug: N-Acetyl-GED-0507-34-LEVO gel 5% — Each patient will apply a fingertip unit of N-Acetyl-GED-0507-34-Levo 5% gel as a thin film, once daily (OD), to the entire facial skin area and the affected skin areas of the trunk accessible for self-application (i.e., shoulders, upper back, and upper anterior chest) for up to 52 consecutive weeks.

SUMMARY:
The clinical trial aims to test the long term safety of a new drug for acne vulgaris. The trial is performed to answer this question "Is it safe to apply the IMP daily for up to 52 weeks?". The trial aims to accurately measure the safety and the effects of the new treatment (N-Acetyl-GED-0507-34-LEVO gel 5%) and to achieve this, patients will be review the drug containing the active ingredient.

Participants will:

* Take drug every day for up to 52 weeks
* Visit the site once every 4 weeks for checkups and tests (where applicable) for the first 3 months of treatment, then visit the site every 13 weeks approximately for checkups and tests (where applicable).
* Record on a diary the daily/weekly applications of the study drug at home, and record any adverse events

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained* * Written informed consent, before any study-related procedure, personally signed and dated by the patient if the patient is ≥ 18 years old or signed and dated by the parents or the legal guardian(s) if the patient is ≥ 9 to < 18 years old. An additional informed assent form must be signed by patient if ≥ 9 to < 18 years old to confirm his willingness to participate in the study. If the patient becomes 18 years of age during the study, the patient must provide written informed consent at that time to continue study participation.
* Sex and age: Male and female patients aged ≥ 9 and < 50 years. Patients who turn 50 during the pivotal study can roll over to the LT study.
* Diagnosis at screening and baseline visits:
* a. Patients affected by facial acne vulgaris with an Investigator's Global Assessment (IGA) score: =1 or 2 for pivotal-naïve* patients not included in pivotal 12 Week treatment studies ≥ 0 for patients completing the 12-Week treatment period according to protocol in the pivotal Phase 3 trials (NAC-GED-0507-ACN-01-23-A and NAC-GED-0507-ACN-01-23-B)
* b. Patients affected by truncal acne (optional criteria) on areas of the trunk (shoulders, upper back and upper anterior chest) accessible for patient's self- application of study medication with a Physician Global Assessment (PGA) severity grade: =1 or 2 for pivotal-naïve* patients not included in the pivotal 12Week treatment studies ≥ 0 and < 4 for patients completing the 12-Week treatment period according to protocol in the pivotal Phase 3 trials (NAC-GED-0507-ACN-01-23-A and NAC-GED-0507-ACN-01-23-B)

  * Pivotal-naïve: Patients not rolling over from NAC-GED-0507-ACN-01-23-A and NAC-GED-0507-ACN-01-23-B. If the pivotal-naïve patient is ≥ 9 and ≤ 14 years old and declined participation to pivotal Phase 3 study, a 12-week period should run before inclusion in the present study. During the 12-week period the patients will be allowed to follow their doctor's instructions regarding treatment of acne.
* Full comprehension Patients and their parents/legal guardian(s) (for < 18 years old patients) can comprehend the whole nature and purpose of the study, including possible risks and side effects, and are able to cooperate with the Investigator and to comply with the requirements of the entire study.
* Contraception and fertility: Women of childbearing potential must be using an effective contraception method during the entire duration of the study. Effective contraception methods are those considered at least "acceptable" according to CTFG Recommendations. A prior stable treatment period is required for the following reliable methods of contraception:

  1. Hormonal oral, implantable, transdermal, or injectable contraceptives must be stable for at least 6 months before the screening visit
  2. A non-hormonal intrauterine device (IUD) must be started at least 2 months before the screening visit.

Exclusion Criteria:

* Acne:

  * Patients with generalized or localized acne forms other than acne vulgaris, e.g., acne conglobata, acne fulminans, acne rosacea, secondary acne (chloracne, drug-induced acne, etc), nodule-cystic acne
  * Patients with acne requiring systemic treatment.
* Beard and facial/body hair, tattoos:

  * Patients with a beard or who intend to grow a beard and/or to perform a facial tattoo during the study
  * Patients with facial hair or facial tattoos that could interfere with study assessments in the investigator's opinion
  * For patients with truncal acne: body hair, tattoos (or who intend to perform them) on the shoulders, upper back or upper anterior chest accessible to self-application of study medication by the patient (evaluable area) that may interfere with the study assessments in the investigator's opinion.
* Skin diseases: Patients with other active skin diseases (e.g., urticaria, atopic dermatitis, sunburn, seborrheic dermatitis, perioral dermatitis, rosacea, skin malignancies) or active skin infections in the facial or truncal region (bacterial, fungal, or viral) or any other facial or truncal disease or condition that might interfere with the evaluation of acne or place the patient at unacceptable risk.
* Allergy: Known or suspected hypersensitivity to any active or inactive ingredient in the study medication. Patients with a history of an allergic reaction or significant sensitivity to the formulations' ingredients.
* Topical therapies: Patients who are currently using, plan to use during the study, or discontinued less than 4 weeks before study baseline the use of prescribed or over-the-counter topical therapies for the treatment of acne, including but not limited to: corticosteroids, antibiotics, azelaic acid, benzoyl peroxide, salicylates, α-hydroxy/glycolic acid, any other topical cosmetic therapy for acne and retinoids on the face/trunk.
* Topical skin care products and procedures: Patients who are currently using, plan to use during the study, or discontinued less than 4 weeks before study baseline the use of products for facial/truncal application containing glycolic or other acids, masks, washes or soaps containing benzoyl peroxide or salicylic acid, non-mild cleansers or moisturizers containing retinol, salicylic or alpha- or beta-hydroxy acids, facial/truncal procedures such as chemical peel, laser treatment, photodynamic therapy, acne surgery, cryodestruction or chemodestruction, x-ray therapy, intralesional steroids, dermabrasion;
* Phototherapy: Patients who are currently using, plan to use during the study, or discontinued less than 4 weeks before study baseline phototherapy for the treatment of acne, including but not limited to: UV-A, UV-B, heliotherapy. Patients who have the need or plan to be exposed to artificial tanning devices or excessive sunlight during the study.
* Systemic therapies: Patients who are currently using, plan to use during the study, or discontinued less than 12 weeks before study baseline the use of systemic therapies for the treatment of acne, including but not limited to: antibiotics, isotretinoin. Other systemic therapy that could affect the patient's acne (i.e., anabolics, lithium, EGRF inhibitors, iodides, systemic corticosteroids - except inhaled corticosteroids or intrathecal corticosteroids - or other immunosuppressants), in the opinion of the investigator.
* Known systemic diseases that can lead to acneiform eruptions:

  1. Increased androgen production.

     1. Adrenal origin: e.g., Cushing's disease, 21-hydroxylase deficiency;
     2. Ovarian origin: e.g., polycystic ovarian syndrome, ovarian hyperthecosis
  2. Cryptococcosis disseminated
  3. Dimorphic fungal infections
  4. Behçet's disease
  5. Systemic lupus erythematosus (SLE).
* Investigative studies: Participation in the evaluation of any other investigational product or device within 24 weeks before study baseline.
* Diseases: Patients with underlying uncontrolled or unstable conditions (including but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal), which, in the Investigator's opinion, could significantly compromise the patient's safety and/or place the patient at an unacceptable risk. Any condition that in the investigator's opinion would make it unsafe for the patient to participate in the study.
* Alcohol and other substance abuse: History of alcohol or other substance abuse within one year before screening.
* Communication: Patient(s) and parents/legal guardian(s) (if applicable) unable to communicate or cooperate with the investigator due to e.g., language problems, impaired cerebral function, impaired mental conditions.
* Reliability: Patients who may be unreliable for the study including patients who are unable to return for the scheduled visits.
* Pregnancy*: Pregnant or breastfeeding women or women of childbearing potential who are planning to become pregnant during the study. *For all female patients of childbearing potential, pregnancy test result must be negative at screening.

Ages: 9 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs, TEAEs, ADRs, SAEs | From enrollment to the end of treatment at 52 weeks
  Incidence of all Adverse Events (AEs), Treatment-Emergent Adverse Events (TEAEs), Adverse Drug Reactions (ADRs), Serious Adverse Events (SAEs) throughout the study; with special attention to local TEAEs concerning the treated facial area (local dermal safety), and systemic TEAEs
Frequency of discontinuation of treatment due to TEAEs | From enrollment to the end of treatment at 52 weeks
Changes from baseline of systolic blood pressure during the study | From enrollment to the end of treatment at 52 weeks
  mmHg
Changes from baseline of diastolic blood pressure during the study | From enrollment to the end of treatment at 52 weeks
  mmHg
Changes from baseline of heart rate during the study | From enrollment to the end of treatment at 52 weeks
  bpm
Physical examination during the study (height) | From enrollment to the end of treatment at 52 weeks
  cm
Change from baseline of local tolerability- Application site signs/symptoms during the study | From enrollment to the end of treatment at 52 weeks
  Local tolerability will be evaluated based on the following signs and symptoms: application site non-lesional erythema, application site exfoliation, and application site dryness, stinging, burning, itching. For each sign/symptom, a severity score will be assigned using a 4-point scale from 0 = absent to 3 = severe. Of note, only a sign/symptom occurring after the first application of study medication that requires additional therapy or discontinuation of treatment or judged from the Investigator as clinically significant will be documented as a TEAE.
Assessment of overall application site irritation over the study duration | From enrollment to the end of treatment at 52 weeks
Physical examination during the study (weight) | From enrollment to the end of treatment at 52 weeks
  kg
Physical examination during the study (BMI) | From enrollment to the end of treatment at 52 weeks
  weight (kg) / [height (m)]²
Changes from baseline of RBC over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement 10E12/L
Changes from baseline of WBC over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement 10E9/L
Changes from baseline of Haematocrit over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement %
Changes from baseline of Haemoglobin over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement g/dl
Changes from baseline of MCV over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement fL
Changes from baseline of MCH over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement pg
Changes from baseline of MCHC over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement g/dL
Changes from baseline of Platelets over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement 10E9/L
Changes from baseline of neutrophils over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement 10E0/L
Changes from baseline of Lymphocytes over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement 10E9/L
Changes from baseline of Monocytes over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement 10E9/L
Changes from baseline of Eosinophils over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement 10E9/L
Changes from baseline of Basophils over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement 10E9/L
Changes from baseline of Differential blood count over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement %
Changes from baseline in AST (GOT) over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement U/L
Changes from baseline in ALT (GPT) over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement U/L
Changes from baseline in Triglycerides over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement mg/dl
Changes from baseline in Total cholesterol over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement mg/dl
Changes from baseline in HDL-C (high-density lipoprotein cholesterol) over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement mg/dl
Changes from baseline in LDL-C (low-density lipoprotein cholesterol) over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement mg/dl
Changes from baseline in Plasma glucose over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement mmol/L
Changes from baseline in HbA1c (glycated haemoglobin) over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement %
Changes from baseline in Insulinemia over the study duration | From enrollment to the end of treatment at 52 weeks
  unit of measurement μU/mL
Changes from baseline in beta-HCG over the study duration | From enrollment to the end of treatment at 52 weeks
  postive or negative

SECONDARY OUTCOMES:
Percentage of patients who have improvement of IGA score at each time point (1, 2 points), vs baseline score (face) | From enrollment to the end of treatment at 52 weeks
The percentage change from baseline in total lesion count (inflammatory plus non-inflammatory) at each time point (face) | From enrollment to the end of treatment at 52 weeks
Absolute change from baseline in total lesion count at each time point (face) | From enrollment to the end of treatment at 52 weeks
Change from baseline in inflammatory lesion count (percentage and absolute), at each time point (face) | From enrollment to the end of treatment at 52 weeks
Change from baseline in non-inflammatory lesion count (percentage and absolute), at each time point. (face) | From enrollment to the end of treatment at 52 weeks
Percentage of patients who have improvement of PGA score at each time point (1, 2 points), vs baseline score | From enrollment to the end of treatment at 52 weeks
The percentage change from baseline in total lesion count (inflammatory plus non-inflammatory) at each time point (trunk) | From enrollment to the end of treatment at 52 weeks
Absolute change from baseline in total lesion count at each time point (trunk) | From enrollment to the end of treatment at 52 weeks
Change from baseline in inflammatory lesion count (percentage and absolute), at each time point (trunk) | From enrollment to the end of treatment at 52 weeks
Change from baseline in non-inflammatory lesion count (percentage and absolute), at each time point. (trunk) | From enrollment to the end of treatment at 52 weeks

OTHER OUTCOMES:
Dermatology Life Quality Index (DLQI) / Children's Dermatology Life Quality Index | From enrollment to the end of treatment at 52 weeks
  C-DLQI for patients from 9 to 16 years old), completed by the patient at V2/Baseline, V5/Wk12 and V8/Wk52 visits (prior to any Investigator assessments to not impact the patient's answers to the quality-of-life questionnaires
Scar Assessment by Scale for Acne Scar Severity (SCAR-S) evaluation at V2/Baseline, V5/Wk12, V6/Wk26, V7/Wk38 and V8/Wk52 visits | From enrollment to the end of treatment at 52 weeks
At selected sites, at V2/Baseline, V5/Wk12 and V8/Wk52 collection of scar 3D photographic documentation will be optional. The area defined for scar assessments is only the face | From enrollment to the end of treatment at 52 weeks

CONTACTS AND LOCATIONS:
Locations (58):
- Italy (18):
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona, AN
  - Azienda USL Toscana Centro, Florence, FI
  - IRCCS Ospedale Policlinico San Martino, Genova, GE
  - Azienda Ospedaliero Universitaria Parma, Parma, PR
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - Azienda Ospedaliera Policlinico Universitario Tor Vergata, Roma, RM
  - I.F.O. Istituti Fisioterapici Ospitalieri, Roma, RM
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS Istituto Di Ricerca E Di Cura A Carattere Scientifico, Bologna
  - Azienda Ospedaliero Universitaria Policlinico G Rodolico San Marco Di Catania, Catania
  - University Hospital Of Ferrara, Ferrara
  - Universita Degli Studi Di Modena E Reggio Emilia, Modena
  - Azienda Ospedaliera Universitaria Federico II Di Napoli, Napoli
  - Azienda Ospedaliera Di Rilievo Nazionale Antonio Cardarelli, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore Della Carita, Novara
  - Azienda Ospedaliera di Padova, Padua
  - Hospital Santa Maria Della Misericordia, Perugia
  - Azienda USL Toscana Centro, Prato
  - Fondazione Luigi Maria Monti, Roma
- Poland (29):
  - Specderm Poznanska Sp. j., Bialystok
  - Vitamed Galaj I Cichomski Sp. j., Bydgoszcz
  - DERMAPOLIS Medical Dermatology Center dr n.med. Edyta Gebska, Chorzów
  - NZOZ Przychodnia Specjalistyczna "A-DERM-SERWIS", Częstochowa
  - Centrum Badan Klinicznych Pi-House Sp. z o.o., Gdansk
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Provita Sp. z o.o., Katowice
  - Silmedic Sp. z o.o., Katowice
  - Vita Longa Sp. z o.o., Katowice
  - Centrum Medyczne Plejady Magdalena Celinska Loewenhoff Michal Zolnowski sp.k., Krakow
  - Jagiellońskie Centrum Innowacji Sp. z o.o., Krakow
  - Amicare Sp. z o.o. S.K., Lodz
  - Dermed Centrum Medyczne Sp. z o.o., Lodz
  - Clinical Best Solutions Sp. z o.o. S.K., Lublin
  - Velocity Nova Sp. z o.o., Lublin
  - St-Inspire Sp. z o.o., Mikołów
  - Twoja Przychodnia Nowosolskie Centrum Medyczne Sp. z o.o., Nowa Sól
  - Etyka Osrodek Badan Klinicznych Tomasz Pesta S.K.A., Olsztyn
  - Labderm Essence Sp. z o.o., Ożarowice
  - Twoja Przychodnia Poznanskie Centrum Medyczne Sp. z o.o., Poznan
  - Uniwersytecki Szpital Kliniczny Im.Fryderyka Chopina W Rzeszowie, Rzeszów
  - Lukmed 2 Sp. z o.o., Siedlce
  - Centrum Zdrowia Dziecka I Rodziny Im. Jana Pawla II W Sosnowcu Sp. z o.o., Sosnowiec
  - Laser Clinic S.C. dr Tomasz Kochanowski dr Andrzej Królicki, Szczecin
  - Twoja Przychodnia Szczecinskie Centrum Medyczne Sp. z o.o., Szczecin
  - Etg Warszawa Sp. z o.o., Warsaw
  - Klinika Ambroziak Sp. z o.o., Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - EMC Instytut Medyczny S.A., Wroclaw
- Spain (11):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Sant Joan De Deu Barcelona Hospital, Esplugues de Llobregat
  - Hospital Universitario Virgen De Las Nieves, Granada
  - Futuremeds Spain S.L., Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario Regional De Malaga, Málaga
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Hospital Quironsalud Infanta Luisa, Seville
  - Futuremeds Spain S.L., Seville
  - Instituto Medico Ricart Valencia S.L., Valencia